CLINICAL TRIAL: NCT03363464
Title: EMPagliflozin compaRative effectIveness and SafEty (EMPRISE) Study Program
Brief Title: Comparative Effectiveness of Empagliflozin in the US
Status: Active, not recruiting | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245.92
Record Dates: First submitted 2017-10-05; First posted 2017-12-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin; Dipeptidyl-Peptidase IV Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients with T2DM initiating empagliflozin: Type 2 diabetes mellitus
  Interventions: Drug: Empagliflozin
- patients with T2DM initiating a DPP-4 inhibitor: dipeptidyl peptidase-4 inhibitor treated patients
  Interventions: Drug: DPP-4 inhibitor
- patients with T2DM initiating a GLP-1 receptor agonist: Glucagon-like peptide-1 receptor agonist treated patients
  Interventions: Drug: GLP-1 receptor agonist

INTERVENTIONS:
Drug: Empagliflozin — Empagliflozin
  Other Names: JARDIANCE, JARDIANZ, GIBTULIO
  Groups: patients with T2DM initiating empagliflozin
Drug: DPP-4 inhibitor — dipeptidyl peptidase-4 inhibitor
  Groups: patients with T2DM initiating a DPP-4 inhibitor
Drug: GLP-1 receptor agonist — Glucagon-like peptide-1 receptor agonist
  Groups: patients with T2DM initiating a GLP-1 receptor agonist

SUMMARY:
Empagliflozin, a sodium glucose co-transporter 2 (SGLT-2) inhibitor, was launched as a treatment for type 2 diabetes mellitus (T2DM) in the U.S. in August 2014. In contrast with several previous cardiovascular outcomes trials, which failed to demonstrate an association with a higher or a lower risk of cardiovascular outcomes associated with members of other recently marketed antidiabetic classes, the EMPA-REG OUTCOME trial has shown that patients at high cardiovascular risk randomized to empagliflozin vs. placebo, were associated with a reduced risk of hospitalization for heart failure, cardiovascular mortality, and all-cause mortality.

However, these and other findings arising from an extensive clinical trial program aimed at evaluating the efficacy and safety profile for empagliflozin have yet to be demonstrated in a non-trial environment. This study aims to investigate the transferability of the effects demonstrated in dedicated randomized clinical studies to a broader population under real world conditions.

ELIGIBILITY:
Inclusion criteria:

* Patients >= 18 years old for Marketscan and Optum, and >=65 years old for Medicare only
* Patients initiating empagliflozin or a DPP-4 inhibitor within the study period. Initiation was defined as no use of SGLT-2 inhibitors (canagliflozin, dapagliflozin, ertugliflozin) or DPP-4 inhibitors in the previous 12 months.
* Restriction to patients with a diagnosis of T2DM (ICD-9 Dx code of 250.x0 or 250.x2; ICD-10 Dx code of E11.x) in the 12 months prior to drug initiation.

Exclusion criteria:

* Patients with missing or ambiguous age or sex information.
* All patients who have less than 12 months of continuous registration in the database prior to initiation of empagliflozin or a DPP-4 inhibitor will be excluded.
* Patients with type 1 diabetes mellitus (T1DM) defined as at least 1 inpatient or outpatient codes in the 12 months prior to drug initiation.
* Secondary diabetes, and gestational diabetes in the 12 months prior to drug initiation
* History of cancer in the 5 years prior to drug initiation
* End-stage renal disease (ESRD) in the 12 months prior to drug initiation
* HIV diagnosis or treatment in the 12 months prior to drug initiation
* Organ transplant in the 12 months prior to drug initiation
* Patients that were in nursing homes in the 12 months prior to drug initiation
* Patients with concomitant SGLT-2 inhibitor and DPP-4 inhibitor initiation will also be excluded.
* Patients initiating more than one DPP-4i on cohort entry date will additionally be excluded Additional exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: T2DM eligible patients in Medicare fee for service, plans A, B, D; United Healthcare (Optum Clinformatics Data Mart); MarketScan (Truven Healthcare Analytics)
Sampling Method: Non-Probability Sample
Enrollment: 230000 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2026-02-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
3-point major adverse cardiovascular events (MACE) | 60 months
  i.e., non-fatal myocardial infarction (MI), non-fatal stroke, or cardiovascular (CV) mortality; as well as each individual component:
  * Hospital admission for MI (for purposes of this individual component, fatal MI is included)
  * Hospital admission for stroke (for purposes of this individual component, fatal stroke is included)
  * CV mortality
Hospitalization for heart failure (specific, based on primary inpatient diagnosis code) | 60 months
Hospitalization for heart failure (broad, based on any inpatient diagnosis code) | 60 months
Modified MACE | 60 months
  i.e., composite of MI, stroke or all-cause mortality
Composite of MI or stroke hospital admission for heart failure | 60 months
All-cause mortality | 60 months

SECONDARY OUTCOMES:
Coronary revascularization procedure | 60 months
Hospitalization for unstable angina | 60 months
Composite of MI, stroke, unstable angina hospitalization or coronary revascularization | 60 months
End-stage renal disease (ESRD) | 60 months
Bone fracture | 60 months
Diabetic ketoacidosis (Inpatient, primary position) | 60 months
Diabetic ketoacidosis (Inpatient, any position) | 60 months
Severe hypoglycemia | 60 months
Urinary tract cancers | 60 months
Lower-limb amputation | 60 months
Acute kidney injury (Inpatient, primary) | 60 months
Acute kidney injury (Inpatient, any position) | 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bringham Women Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Patorno E, Pawar A, Franklin JM, Najafzadeh M, Deruaz-Luyet A, Brodovicz KG, Sambevski S, Bessette LG, Santiago Ortiz AJ, Kulldorff M, Schneeweiss S. Empagliflozin and the Risk of Heart Failure Hospitalization in Routine Clinical Care. Circulation. 2019 Jun 18;139(25):2822-2830. doi: 10.1161/CIRCULATIONAHA.118.039177. Epub 2019 Apr 8. PMID 30955357
- See also: Related Info — https://www.mystudywindow.com